CLINICAL TRIAL: NCT02602977
Title: the Influence of Remote Ischemic Preconditioning on Inflammation During Human Endotoxemia, a Pilot Proof-of-principle Study
Brief Title: the Influence of Remote Ischemic Preconditioning on Inflammation During Human Endotoxemia
Acronym: RISPENDO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RISPENDO
Record Dates: First submitted 2015-09-30; First posted 2015-11-11 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Autoimmune Diseases; Infection
Keywords: inflammation; remote ischemic preconditioning
MeSH Terms: conditions — Autoimmune Diseases; Infections; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- multiple-dose RIPC (Experimental): Multiple-dose Remote Ischemic Preconditioning. A group of 10 subjects that will receive 4 cycles of remote ischemic preconditioning of the upper limb per day in the 7 consecutive days before the endotoxemia experiment. The last dose will be applied 40 minutes before LPS administration.
  Interventions: Other: Multiple-dose Remote Ischemic Preconditioning; Biological: LPS infusion
- single-dose RIPC (Experimental): Single-dose Remote Ischemic Preconditioning. A group of 10 subjects that will receive a single RIPC dose, starting 40 minutes before LPS administration.
  Interventions: Other: Single-dose Remote Ischemic Preconditioning; Biological: LPS infusion
- control group (Active Comparator): Only LPS infusion. A group of 10 subjects that will be administered LPS without RIPC.
  Interventions: Biological: LPS infusion

INTERVENTIONS:
Other: Multiple-dose Remote Ischemic Preconditioning — A blood-pressure cuff with handheld rubber inflation balloon and manometer is placed on the non-dominant arm of the subject. The cuff will be placed proximally from the elbow with the most proximal part of the cuff placed in the armpit. The cuff will be inflated to 250 mmHg after which a 5 minute countdown is started. After 5 minutes the pressure is released and the 5 minute countdown for reperfusion is started. This concludes one cycle out of a total of four.
  1 "RIPC-dose" consists of 4 cycles of 5 minute ischemia followed by 5 minute reperfusion as described above.
  Multiple-dose RIPC consists of a daily dose of 1 RIPC as described above for 7 consecutive days.
  Other Names: RIPC
  Arms: multiple-dose RIPC
Other: Single-dose Remote Ischemic Preconditioning — A blood-pressure cuff with handheld rubber inflation balloon and manometer is placed on the non-dominant arm of the subject. The cuff will be placed proximally from the elbow with the most proximal part of the cuff placed in the armpit. The cuff will be inflated to 250 mmHg after which a 5 minute countdown is started. After 5 minutes the pressure is released and the 5 minute countdown for reperfusion is started. This concludes one cycle out of a total of four.
  1 "RIPC-dose" consists of 4 cycles of 5 minute ischemia followed by 5 minute reperfusion as described above.
  Single-dose RIPC consists of 1 dose of RIPC as described above
  Other Names: RIPC
  Arms: single-dose RIPC
Biological: LPS infusion — To achieve a controlled inflammatory state, 30 subjects (multiple-dose RIPC group [n=10], single-dose RIPC group [n=10] and control group [n=10]) will receive LPS intravenously. The LPS at a dose of 2 ng/kg iv will be injected in 1 minute.
  Other Names: human endotoxemia

SUMMARY:
In a wide range of auto-inflammatory and infectious diseases attenuation of the immune response could be beneficial. Remote ischemic preconditioning (RIPC) has been identified as a means of protecting patients undergoing cardiac surgery from perioperative myocardial ischemic damage. This protection can be divided in a 'first window of protection' directly after preconditioning and a 'second window' that protects patients 12-48 hour after preconditioning. Repeated RIPC might have additional value, possibly by combining beneficial effects of the first and second windows of protection. The mechanisms behind these effects are under investigation, but attenuation of the inflammatory response is a major candidate. However, this has not yet been demonstrated in the setting of systemic inflammation in humans in vivo. This study aims to investigate the effects of (repeated) ischemic preconditioning on inflammation during human endotoxemia.

DETAILED DESCRIPTION:
Although the immune system is essential to survival, a variety of diseases originate from inappropriate or excessive activation of the immune response. Examples include a wide range of auto-inflammatory disease, infectious diseases such as sepsis, but also after major surgery like cardiac artery bypass grafting, after radiation therapy in the treatment of cancer, or following organ transplantation. In these instances, attenuation of the immune response could be beneficial.

The concept of ischemic preconditioning (IPC) was first described in the 1980's. Murry and colleagues showed a protective effect of preconditioning the heart with 4 cycles of 5-minute long ischemia on the extent of myocardial infarction in dog hearts. Follow-up animal studies showed the same protective effects on the heart by introducing the cycles of ischemia to distant, or 'remote', organs like the kidney or the gut. Furthermore, this principle of 'remote ischemic preconditioning' (RIPC) was also shown to be effective in humans when using a tourniquet to temporary cut off blood supply to one of the limbs, either an arm or a leg. As such, RIPC has been identified as a cheap and easy method of protecting patients undergoing elective CABG surgery from perioperative myocardial ischemic damage. In recent studies, two different timeframes in which RIPC exerts its protective effects have been identified. The classical or 'early window of protection' protects in the 1-2 hour after the RIPC stimulus while a 'second window of protection' is evident 12-24 hours after RIPC and lasts for 48-72 hours. Multiple-dose RIPC may be of additional value, as 7 daily doses of RIPC in humans resulted in protection of endothelial dysfunction, with both the local and remote beneficial effects lasting for up to 8 days after the last RIPC dose. This could be due to additive or synergistic effects of combining the first and second windows of protection.

The mechanisms behind the observed protective effects are however still subject of investigation. Several have been put forward, of which attenuation of the inflammatory response is a major candidate.

For instance, recent animal work has shown that RIPC results in downregulation of pro-inflammatory cytokines such as TNF-α and IL-6 and upregulation of anti-inflammatory cytokines such as IL-10. In support of the latter, the cardioprotective effects of RIPC were absent in IL-10 knockout mice or in wild-type mice treated with a monoclonal antibody against the IL-10 receptor. Hypoxia-inducible factor (HIF) has been shown to be a major contributor to this RIPC-induced IL-10 response.

Adenosine appears to be a major determinant of the anti-inflammatory and tissue-protective effects of RIPC. In a in vivo forearm model, adenosine and ischemic preconditioning both resulted in the same reduction in ischemia-reperfusion injury. Also, administration of exogenous adenosine can mimic the protective effects of IPC, and antagonizing the adenosine receptor with caffeine blocks the protective effects of RIPC and augments the anti-inflammatory IL-10 response to lipopolysaccharide (LPS). Interestingly, one of the pathways in which ischemia-reperfusion can increase adenosine levels is through upregulation of CD73, which is dependent on the aforementioned HIF.

Another possible mechanism behind the anti-inflammatory effects of RIPC is release of Toll-like receptor (TLR) ligands, which in turn induce an endotoxin tolerance-like state. Endotoxin tolerance is a refractory state of the immune system after challenge with the TLR4 ligand LPS, characterized by diminished cytokine production upon a subsequent LPS challenge. However, induction of endotoxin tolerance was found to occur not only after LPS challenge but also using other TLR(4)-ligands, so-called 'cross-tolerance'. A possible candidate to induce tolerance in RIPC is heat shock protein 70 (HSP70), as extracellular HSP70 has been shown to induce tolerance to LPS in monocytes in vitro. Furthermore, in rats receiving ischemic preconditioning of the lower extremity, HSP70 expression was increased in the spinal cord and myocardium, and HSP70 upregulation was found in cardiomyocytes after RIPC in infants undergoing cardiac surgery. However, other, yet unidentified TLR ligands could also be involved.

From the abovementioned studies, it appears that RIPC exerts significant effects on the immune response. However, this has not yet been demonstrated in the setting of systemic inflammation in humans in vivo. Furthermore, the mechanisms behind the putative anti-inflammatory effects and possible additive or synergistic effects of repeated RIPC (thereby combining both the first and second windows of protection) are unknown as well. This study aims to investigate the effects of (repeated) ischemic preconditioning during human endotoxemia, a standardized controlled model of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in this trial
* Male subjects aged 18 to 35 years inclusive
* Healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram and clinical laboratory parameters

Exclusion Criteria:

* Use of any medication
* Smoking
* Use of recreational drugs within 21 days prior to endotoxemia experiment day
* Use of caffeine or alcohol within 1 day prior to endotoxemia experiment day
* Previous participation in a trial where LPS was administered
* Surgery or trauma with significant blood loss or blood donation within 3 months prior to endotoxemia experiment day
* Participation in another clinical trial within 3 months prior to endotoxemia experiment day
* History, signs, or symptoms of cardiovascular disease
* History of frequent vaso-vagal collapse or of orthostatic hypotension
* History of atrial or ventricular arrhythmia
* Hypertension (RR systolic >160 or RR diastolic >90)
* Hypotension (RR systolic <100 or RR diastolic <50)
* Conduction abnormalities on the ECG consisting of a 1st degree atrioventricular block or a complex bundle branch block
* Renal impairment: plasma creatinine >120 µmol/L
* Liver function abnormality: alkaline phosphatase>230 U/L and/or ALT>90 U/L
* History of asthma
* Obvious disease associated with immune deficiency
* CRP > 20 mg/L, WBC > 12x109/L, or clinically significant acute illness, including infections, within 4 weeks before endotoxemia day

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Plasma TNF-α concentration following LPS administration | 1 day
  The primary study parameter is the difference in circulating TNF-α concentration over time between the multiple-dose (7 days) RIPC group and the control group.

SECONDARY OUTCOMES:
circulating cytokines (including but not limited to IL-6, IL-10, IL-1RA) | 1 day
Hemodynamic parameters | 1 day
  blood pressure, heart frequency, respiratory frequency
body temperature | 1 day
subjective symptom scores | 1 day
  The subject is asked to score the severity of experienced symptoms every 30 minutes throughout the experiment. Symptom are scored on a scale ranging from 0, (symptom not present) to 5 (worst ever experienced).
kidney injury markers in urine - TIMP2*IGFBP7 | 1 day
  TIMP2*IGFBP7 (expressed in ng/ml^2) is a combined marker that is measured using the NephroCheck Test (Astute Medical, San Diego, CA, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Jelle Zwaag, MSc, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Intensive Care, Nijmegen, Netherlands

REFERENCES:
- [Derived] Zwaag J, Beunders R, Warle MC, Kellum JA, Riksen NP, Pickkers P, Kox M. Remote ischaemic preconditioning does not modulate the systemic inflammatory response or renal tubular stress biomarkers after endotoxaemia in healthy human volunteers: a single-centre, mechanistic, randomised controlled trial. Br J Anaesth. 2019 Aug;123(2):177-185. doi: 10.1016/j.bja.2019.03.037. Epub 2019 May 10. PMID 31084985